CLINICAL TRIAL: NCT00977639
Title: Evaluation of Pathwork Tissue of Origin (TOO) Test for Human Malignancies
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: James L Zehnder, Stanford University School of Medicine
Other Study IDs: SU-03072008-1032; 98301; VAR0029
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a tissue biopsy specimen

INTERVENTIONS:
Procedure: Pathwork TOO test

SUMMARY:
The pathworks tissue of origin test is a microarray-based test with the goal of identifying the tissue of origin in patients with metastatic tumors of unknown primary site.

ELIGIBILITY:
Inclusion Criteria:1 Subjects must be at least 18 years old. The TOO test is designed to determine the tissue of origin of common adult malignancies. There are no gender/ethnic restrictions.

2 Patients with a diagnosis of malignancy established by pathologic review of H&E staining of tumor biopsy or tumor resection without definitive determination of tissue of origin as assessed by the PI. Samples must have been obtained within three months of enrollment, or the patient must still be under active evaluation for tissue of origin at the time of enrollment. There are no limitations on prior therapy and time from last prior therapy.

3 Ability to understand and the willingness to sign a written informed consent document. Exclusion Criteria:1 Patients under the age of 18 are excluded. There are no exclusions based on gender/ethnicity.

2 There are no exclusion requirements due to co-morbid disease or incurrent illness, as needed.

3 Pregnancy or nursing participants will not be excluded from the study.

4 Patients with a diagnosis of leukemia including acute myelogenous leukemia, acute lymphocytic leukemia, hairy cell leukemia, chronic myelogenous leukemia and chronic lymphocytic leukemia are excluded from enrollment on this study. The TOO test does not cover these diagnoses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of malignancy
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Zehnder, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States